CLINICAL TRIAL: NCT01056081
Title: Inspiratory Muscle Training for Patients With Chronic Obstructive Pulmonary Disease Undergoing a Pulmonary Rehabilitation Program
Brief Title: Inspiratory Muscle Training in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Faculdade Evangelica do Parana (Other)
Responsible Party: Silvia Valderramas, Faculdade Evangélica do Paraná
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FEPAR 1768
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2006-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; inspiratory muscles; diaphragm
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inspiratory muscle training (Experimental): The training was performed using a threshold inspiratory muscle trainer (Respironics HealthScan, Inc, Cedar Grove, New York, USA).
  The patients performed the IMT training in a seated position, with the upper limbs supported. The total duration of the respiratory training was 30 minutes, with sequences of three minutes of training followed by pauses of two minutes. The initial load was equivalent to 30% of the individual's MIP. This load was progressively increased over the first four weeks, according to the patients' tolerance, to reach 60% of the MIP. This level was then maintained until the end of the training.
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — The training was performed using a threshold inspiratory muscle trainer (Respironics HealthScan, Inc, Cedar Grove, New York, USA).
  The patients performed the IMT training in a seated position, with the upper limbs supported. The total duration of the respiratory training was 30 minutes, with sequences of three minutes of training followed by pauses of two minutes. The initial load was equivalent to 30% of the individual's MIP. This load was progressively increased over the first four weeks, according to the patients' tolerance, to reach 60% of the MIP. This level was then maintained until the end of the training.
  Other Names: IMT

SUMMARY:
Uncertainty persists regarding the usefulness of incorporating inspiratory muscle training (IMT) in pulmonary rehabilitation programs for patients with chronic obstructive pulmonary disease. In this study the investigators investigate whether IMT associated with exercise training would be better than exercise training alone, with regard to exercise capacity, inspiratory muscle strength and dyspnea.

DETAILED DESCRIPTION:
Study design: A double-blind parallel controlled trial Setting: outpatient clinic Inclusion criteria: Subjects between 40 and 75 years of age referred by a physician to the Pulmonary Rehabilitation Program, with a clinical and spirometric diagnosis of moderate to severe COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD).

Outcome measurements: Inspiratory muscle strength (using maximal inspiratory pressure, MIP), exercise capacity (using six-minute walk test) and dyspnea were measured.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical and spirometric diagnosis of moderate to severe COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD)
* In a stable condition (without exacerbations or infections for at least a month)
* Had to be former smokers (> 6 months without smoking)
* subjects referred by a physician to the Pulmonary Rehabilitation Program

Exclusion Criteria:

* Subjects with a known history of asthma, or severe and/or unstable heart disease or any other pathological condition that could impair their physical activities

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Inspiratory muscle strength | 8 weeks

SECONDARY OUTCOMES:
Exercise capacity | 8 weeks
Dyspnea | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R Valderramas, PhD, Study Chair — Evangelical Faculty of Paraná